CLINICAL TRIAL: NCT03085784
Title: Intravitreal Aflibercept Injection (IAI) for Radiation Retinopathy Trial (ARRT)
Brief Title: Intravitreal Aflibercept Injection for Radiation Retinopathy Trial
Acronym: ARRT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amy C Schefler, MD (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Amy C Schefler, MD, Principal Investigator, Greater Houston Retina Research
Organization: Greater Houston Retina Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARRT
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Radiation Retinopathy
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Loading Dose (Experimental): 20 Patients will receive 4, 2 mg IVT Aflibercept (IAI) a month apart, screening/baseline, weeks 4, 8, & 12. At week 12, patient will be followed & treated per treat & extend protocol.
  Treat & Extend Protocol entails patients being extended as long as:
  * Absence of retinal fluid (resolution of intraretinal & subretinal fluid on SD-OCT; Small intraretinal cysts that don't distort foveal contour on SD-OCT are acceptable & can be considered "dry".) AND
  * < 5 ETDRS letter loss from previous visit, due to new or persistent retinal edema.
  Each extension will be 2 weeks in duration beyond the initial 4-week interval. If the extension criteria are not met on a follow-up visit, treatment interval will be reduced by 2 weeks. Follow up interval will continue to be reduced by 2 weeks until the extension criteria are met or a 4-week interval is reached.
  Interventions: Drug: Aflibercept
- Treat and Extend (Experimental): 20 Patients will receive 2 mg IVT Aflibercept (IAI) at screening/baseline followed by a visit at week 4. At week 4, patient will be treated & followed per the treat & extend protocol.
  Treat & Extend Protocol entails patients being extended as long as:
  * Absence of retinal fluid (resolution of intraretinal & subretinal fluid on SD-OCT; Small intraretinal cysts that don't distort foveal contour on SD-OCT are acceptable & can be considered "dry".) AND
  * < 5 ETDRS letter loss from previous visit, due to new or persistent retinal edema.
  Each extension will be 2 weeks in duration beyond the initial 4-week interval. If the extension criteria are not met on a follow-up visit, treatment interval will be reduced by 2 weeks. Follow up interval will continue to be reduced by 2 weeks until the extension criteria are met or a 4-week interval is reached.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — The investigational product is intravitreal aflibercept injection (IAI), which will be supplied by Regeneron Pharmaceuticals, Inc. in sterile vials for intravitreal (IVT) injection. The study duration will be 52 weeks. Vials of drug must be used (defined as entered with needle) only once. All drug supplies are to be kept under recommended storage conditions. The injection volume will be 50μL (0.05 mL) and will be administered to the patients by IVT injection.
  Other Names: Eylea

SUMMARY:
The ARRT trial will assess the safety and efficacy of 2mg aflibercept for the treatment of radiation retinopathy, including maculopathy and optic neuropathy over 52 weeks.

DETAILED DESCRIPTION:
Approximately 40 eyes will be randomized (1:1 ratio) into either Group 1 or Group 2. Slit lamp exam and Indirect ophthalmoscopy will be performed at every study visit, where retinopathy level will be assessed. SD-OCT will be performed at each visit. Fluorescein angiogram will be performed at screen, week 26 and week 52. All other imaging studies will be standard of care at the discretion of the investigator.

This trial will compare the results of 2 groups, with different treatment intervals, to assess the safety of intravitreal Aflibercept injections (IAI) for the treatment of radiation retinopathy. Patients in each group will be followed for a total of 52 weeks.

Group 1: 15 Patients will receive a loading dose of 3 IAI. They will receive 2 mg IAI at screening/baseline, week 4, week 8, and week 12. A follow-up visit will occur at week 12. If the extension criteria are met, the patient will be extended by 2 weeks. The patient will continue to be followed per the treat and extend protocol described below.

Group 2: Patients will not receive a loading dose. They will receive 2 mg IAI at screening/baseline followed by a visit at week 4. At week 4, if the extension criteria are met, the patient will be extended by 2 weeks. The patient will continue to be followed per the treat and extend protocol described below.

Treat & Extend Protocol Patients can be extended as long as they meet the following criteria -

* Absence of retinal fluid (resolution of intraretinal and subretinal fluid on SD-OCT; Small intraretinal cysts that do not distort foveal contour on SD-OCT are acceptable and can be considered "dry".) AND
* Less than 5 ETDRS letter loss from previous visit due to new or persistent retinal edema.

IAI will be rendered at every visit (treatment at the week 26 mandatory visit will be administered based on the treat and extend status), no earlier than 4 days before the target date and no later than 4 days after the target date. Each extension will be 2 weeks in duration beyond the initial 4-week interval. If the extension criteria are not met on a follow-up visit, the treatment interval will be reduced by 2 weeks. Follow up interval will continue to be reduced by 2 weeks until the extension criteria are met or a 4-week interval is reached.

All patients will have a mandatory study visit at Week 52 (final study visit). No study treatment will be administered after week 50 or at a study termination visit. If a patient receives treatment after week 48, they will return 4 weeks after the last clinic visit for the final study visit (instead of at week 52).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years of age
2. Clinically identifiable radiation retinopathy with evidence of fluid on SD-OCT causing vision loss in the study eye
3. Undergone either ocular or orbital radiation for any primary ocular or orbital cancer within clinical evidence of having radiation retinopathy
4. Willing and able to comply with clinic visits and study-related procedures
5. Provide signed informed consent

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from the study:

1. Metastatic cancer or any active primary cancer, at time of enrollment
2. Prior treatment with anti VEGF in the study within 60 days of screen in the study eye
3. Prior intravitreal or subconjunctival treatment with cortical steroids within 90 days of screen in the study eye
4. Macular ischemia (defined as greater than 5 disc areas), as assessed by the investigator
5. Media opacity obscuring a view of the fundus or any other reason for vision loss other than radiation retinopathy.
6. Evidence of infectious ocular infection, in the study eye, at time of screening
7. Pregnant or breast-feeding women
8. Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception start of the first treatment, during the study, and for at least 3 months after the last dose. Adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly.

   * Contraception is not required for men with documented vasectomy. **Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of childbearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-07-05 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Safety of intravitreal Aflibercept for the treatment of radiation retinopathy - Assessed by incidence of adverse events. | 52 Weeks
  The primary objective of the study is to assess the safety of 2 mg intravitreal Aflibercept injections (IAI) for the treatment of radiation retinopathy including maculopathy and optic neuropathy. Assessed by incidence of adverse events.

SECONDARY OUTCOMES:
Resolution of macular edema (CRT) | 52 Weeks
  Resolution of macular edema as measured by mean change in central retinal thickness
Resolution of macular edema (% dry) | 52 Weeks
  Resolution of macular edema as measured by % of patients who achieve a dry macula
Stabilization and improvement in visual acuity | 52 Weeks
  Stabilization and improvement in visual acuity as measured by the mean change in Early Treatment Diabetic Retinopathy Study best-corrected visual acuity
Dosing frequency of intravitreal aflibercept injections | 52 Weeks
  Dosing frequency of IAI as measured by number of injections
Incidence of neovascularization, vitreous hemorrhage, and need for vitrectomy | 52 Weeks
  Percentage of patients avoiding the development of increased neovascularization, vitreous hemorrhage, and need for vitrectomy
Resolution of retinal hemorrhage, retinal exudates, optic disc edema, and capillary non-perfusion | 52 Weeks
  Percentage of patients with resolution of retinal hemorrhages, retinal exudates, optic disc edema, capillary non-perfusion

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Schefler, MD, Principal Investigator — Retina Consultants Houston
Locations (3):
- United States (3):
  - Retina Consultants of Houston/Texas Medical Center, Houston, Texas
  - Retina Consultants of Houston, Katy, Texas
  - Retina Consultants of Houston/The Woodlands, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jampol LM, Moy CS, Murray TG, Reynolds SM, Albert DM, Schachat AP, Diddie KR, Engstrom RE Jr, Finger PT, Hovland KR, Joffe L, Olsen KR, Wells CG; Collaborative Ocular Melanoma Study Group (COMS Group). The COMS randomized trial of iodine 125 brachytherapy for choroidal melanoma: IV. Local treatment failure and enucleation in the first 5 years after brachytherapy. COMS report no. 19. Ophthalmology. 2002 Dec;109(12):2197-206. doi: 10.1016/s0161-6420(02)01277-0. PMID 12466159
- [Background] Melia BM, Abramson DH, Albert DM, Boldt HC, Earle JD, Hanson WF, Montague P, Moy CS, Schachat AP, Simpson ER, Straatsma BR, Vine AK, Weingeist TA; Collaborative Ocular Melanoma Study Group. Collaborative ocular melanoma study (COMS) randomized trial of I-125 brachytherapy for medium choroidal melanoma. I. Visual acuity after 3 years COMS report no. 16. Ophthalmology. 2001 Feb;108(2):348-66. doi: 10.1016/s0161-6420(00)00526-1. PMID 11158813
- [Background] Gunduz K, Shields CL, Shields JA, Cater J, Freire JE, Brady LW. Radiation retinopathy following plaque radiotherapy for posterior uveal melanoma. Arch Ophthalmol. 1999 May;117(5):609-14. doi: 10.1001/archopht.117.5.609. PMID 10326957
- [Background] Finger PT, Chin KJ. High-dose (2.0 mg) intravitreal ranibizumab for recalcitrant radiation retinopathy. Eur J Ophthalmol. 2013 Nov-Dec;23(6):850-6. doi: 10.5301/ejo.5000333. Epub 2013 Jun 28. PMID 23813109
- [Background] Finger PT, Chin KJ. Intravitreous ranibizumab (lucentis) for radiation maculopathy. Arch Ophthalmol. 2010 Feb;128(2):249-52. doi: 10.1001/archophthalmol.2009.376. No abstract available. PMID 20142553
- [Background] Finger PT, Chin KJ. Antivascular endothelial growth factor bevacizumab for radiation optic neuropathy: secondary to plaque radiotherapy. Int J Radiat Oncol Biol Phys. 2012 Feb 1;82(2):789-98. doi: 10.1016/j.ijrobp.2010.11.075. Epub 2011 Jan 27. PMID 21277107
- [Background] Finger PT, Mukkamala SK. Intravitreal anti-VEGF bevacizumab (Avastin) for external beam related radiation retinopathy. Eur J Ophthalmol. 2011 Jul-Aug;21(4):446-51. doi: 10.5301/EJO.2011.6213. PMID 21218391
- [Background] Mason JO 3rd, Albert MA Jr, Persaud TO, Vail RS. Intravitreal bevacizumab treatment for radiation macular edema after plaque radiotherapy for choroidal melanoma. Retina. 2007 Sep;27(7):903-7. doi: 10.1097/IAE.0b013e31806e6042. PMID 17891015
- [Background] Finger PT. Radiation retinopathy is treatable with anti-vascular endothelial growth factor bevacizumab (Avastin). Int J Radiat Oncol Biol Phys. 2008 Mar 15;70(4):974-7. doi: 10.1016/j.ijrobp.2007.11.045. PMID 18313522
- [Background] Finger PT, Chin K. Anti-vascular endothelial growth factor bevacizumab (avastin) for radiation retinopathy. Arch Ophthalmol. 2007 Jun;125(6):751-6. doi: 10.1001/archopht.125.6.751. PMID 17562985
- [Background] Gupta A, Muecke JS. Treatment of radiation maculopathy with intravitreal injection of bevacizumab (Avastin). Retina. 2008 Jul-Aug;28(7):964-8. doi: 10.1097/IAE.0b013e3181706302. PMID 18698298
- [Background] Kim IK, Lane AM, Jain P, Awh C, Gragoudas ES. Ranibizumab for the Prevention of Radiation Complications in Patients Treated With Proton Beam Irradiation for Choroidal Melanoma. Trans Am Ophthalmol Soc. 2016 Aug;114:T2. PMID 27630373

DOCUMENTS (2):
  • Informed Consent Form (2017-05-03): https://cdn.clinicaltrials.gov/large-docs/84/NCT03085784/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT03085784/Prot_SAP_001.pdf